CLINICAL TRIAL: NCT01312519
Title: A Trial of the Vidacare Powered Bone Marrow Aspiration and Core Biopsy Systems (OnControl by Vidacare) Compared to Traditional Manual Devices
Brief Title: Powered Bone Marrow Aspiration and Core Biopsy System Compared to Manual Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Organization: Teleflex (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-04
Record Dates: First submitted 2010-11-03; First posted 2011-03-10 (Estimated); Results first posted 2013-07-23 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2013-07

CONDITIONS: Bone Marrow Biopsy Procedures
Keywords: Bone marrow biopsy of iliac crest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual bone marrow sampling device (Active Comparator): Hollow needle with a t-shaped handle manually pushed into the bone for the purpose of bone marrow aspiration and core biopsy collection. Manual Bone Marrow Sampling Device.
  Interventions: Device: Manual bone marrow sampling device
- OnControl Bone Marrow System (Active Comparator): Battery powered device used for insertion of a single lumen catheter into the intraosseous space of the adult iliac crest. OnControl Bone Marrow Biopsy and Aspiration System.
  Interventions: Device: OnControl Bone Marrow Biopsy and Aspiration System

INTERVENTIONS:
Device: OnControl Bone Marrow Biopsy and Aspiration System — Battery powered device used for insertion of a single lumen catheter into the intraosseous space of the adult iliac crest for the purpose of aspiration and core biopsy collection.
  Other Names: OnControl; Powered Biopsy Device
  Arms: OnControl Bone Marrow System
Device: Manual bone marrow sampling device — Hollow needle with a t-shaped handle that is pushed into the bone for the purpose of collecting bone marrow aspiration and core biopsy samples.
  Other Names: Jamshidi; Manual biopsy needle
  Arms: Manual bone marrow sampling device

SUMMARY:
This is a randomized study evaluating use of a powered bone marrow biopsy and aspiration system (OnControl by Vidacare) compared to traditional manual devices. The hypothesis is that the powered system will reduce the level of patient pain during the aspiration and core biopsy procedures and the amount of time needed to perform the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18
* Patients that require core biopsy alone, or core biopsy and bone marrow aspiration

Exclusion Criteria:

* Imprisoned
* Pregnant
* Cognitively impaired
* Requiring english language translation other than Spanish
* Patients with one or more conditions precluding bone marrow core biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Philbeck, PhD, Study Director — Vidacare Corporation
Locations (2):
- Cancer Therapy and Research Center, San Antonio, Texas, United States
- Hospital General Universitario Gregorio Maranon, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients 18 years of age requiring bone marrow aspiration and biopsy as part of routine care were considered eligible for the study.
Pre-assignment Details: No pre-assisgnment details.
Groups:
- Manual Bone Marrow Sampling Device: hollow needle with a t-shaped handle manually pushed into the bone for the purpose of bone marrow aspiration and core biopsy collection.
- OnControl Bone Marrow System: Battery powered device used for insertion of a single lumen catheter into the intraosseous space of the adult iliac crest.
Period: Overall Study
Arm/Group | Manual Bone Marrow Sampling Device | OnControl Bone Marrow System
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Bone Marrow Sampling Device | OnControl Bone Marrow System | Total
Number analyzed (Participants) | 26 | 24 | 100
Age, Categorical [Count of Participants; unit: Participants]
  number analyzed (Participants) | 26 | 24 | 50
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years]
  number analyzed (Participants) | 26 | 24 | 50
  (all) | 59 (17) | 53 (19.0) | 56.0 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 26 | 24 | 50
  Female | 12 | 9 | 21
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States: number analyzed (Participants) | 26 | 24 | 50
  United States | 12 | 18 | 30
  Spain: number analyzed (Participants) | 26 | 24 | 50
  Spain | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Level of Pain During Procedure
Description: Subjects were asked to rate the level of pain they experienced during the procedure for needle insertion, following penetration of the cortex. A 0 to 10 pain scale was used where 0=no pain and 10= worst possible pain.
Time Frame: Day 1 during the needle insertion
Population: as per protocol, 50 patients were enrolled in the study and randomized to the manual bone marrow sampling device or the battery powered device.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manual bone marrow sampling device | OnControl Bone Marrow System
Number analyzed (Participants) | 26 | 24
units on a scale | 3.8 (3.0) | 3.2 (2.2)

2. Secondary Outcome: Time Necessary to Perform the Bone Marrow Procedure
Description: The time necessary to perform the procedure was measured as follows: Time started once the needle and skin came into contact and time stopped once the sample was collected and the needle was removed from the patient.
Time Frame: Day 1 needle insertion through needle removal
Population: Per protocol, 50 patients were enrolled in the study and randomized to the manual bone marrow sampling device or the battery powered device.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Manual bone marrow sampling device | OnControl Bone Marrow System
Number analyzed (Participants) | 26 | 24
seconds | 224.1 (79.0) | 100.0 (72.8)

ADVERSE EVENTS:
Arm/Group | Manual Bone Marrow Sampling Device | OnControl Bone Marrow System
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less